CLINICAL TRIAL: NCT00744159
Title: Prospective Comparative Study of Immunological Benefit Between Laparoscopic Colectomy and Open Colectomy
Brief Title: Prospective Comparison of Immunological Benefit of Laparoscopic Colectomy
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Woo Yong Lee/Associate Professor, Department of Surgery, Samsung Medical Center, Samsugn Medical Center
Other Study IDs: IRB 2005-08-041; #CRS-106-14-1
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Immunity
Keywords: colon cancer; laparoscopic colorectal surgery; cellular immunity; HLA-DR expression on monocyte
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OC: Open colorectal resection
- LC: Laparoscopic colorectal resection

SUMMARY:
This study aimed to clarify existence of immunological benefit of laparoscopic colon cancer surgery compared to open colon surgery.

DETAILED DESCRIPTION:
Patients with clinical stage Ⅲ left colon and upper rectal cancer were prospectively assigned to undergo LC (n=35) or OC (n=39). Factors related to cellular immunity of host (total lymphocyte count, CD4 lymphocyte, CD8 lymphocyte, CD4/CD8 ratio, HLA-DR expression on monocyte (mHLA-DR)) were examined preoperatively, on the 1st day of operation (POD1) and the 5th day of operation (POD5).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven of colon cancer
* Preoperatively suspected as clinical stage III colon cancer
* Lesion located Descending colon, sigmoid colon and upper rectal cancer

Exclusion Criteria:

* Could not perform curative resection
* Intestinal obstruction, perforation, intra-abdominal abscess
* Severe medical illness
* Immunopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital based cohort
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Immune factors | post OP 5th day

SECONDARY OUTCOMES:
Post-operative complications | POD 7th days

CONTACTS AND LOCATIONS:
Overall Officials: Woo Yong Lee, MD,PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Department of surgery, Seoul, South Korea